CLINICAL TRIAL: NCT06328751
Title: Study With Cancer Patients at the CECON Foundation's Pain Therapy and Palliative Care Service: Meditation With Immersive Virtual Reality for Pain Relief
Brief Title: Meditation With Virtual Reality for Cancer Pain Relief in the Pain Therapy and Palliative Care Service
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Santos Montarroyos (Network)
Collaborators: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Emily Santos Montarroyos, physician, FUNDAÇÃO CENTRO DE CONTROLE DE ONCOLOGIA DO ESTADO DO AMAZONAS
Organization: FUNDAÇÃO CENTRO DE CONTROLE DE ONCOLOGIA DO ESTADO DO AMAZONAS (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 76043823.0.0000.0004
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cancer Pain; Quality of Life; Palliative Medicine
Keywords: Meditation; Cancer Pain; Quality of Life; Virtual Reality
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, experimental, longitudinal, randomized controlled trial (RCT), carried out in three stages.
Who Masked: Participant
Masking Description: Randomization will be carried out using a specific application called Randomizer ® for Clinical Trial Lite, which is a secure and validated application that works with encrypted network traffic using Transport Layer Security (TLS), a strong encryption. There will be 3 groups which will be divided into the Case Group, the Active Control Group and the Passive Control Group. Each patient will be seen individually wearing a Samsung® smartwatch and will not know about the other patients' meditation. The case group will watch a 7-minute immersive virtual reality video of mindfulness meditation with image and sound in the Oncology Control Center Foundation (FCECON) office, using Samsung® gear VR virtual reality glasses. The active control group will watch a 7-minute mindfulness meditation video presented via cell phone with image and sound at the office. The passive control group will perform breathing exercises based on the healthcare professional's instructions for 4 minutes in the office.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Case Group (Experimental): The case group will watch a 7-minute immersive virtual reality video of mindfulness meditation with image and sound in the office of the Oncology Control Center Foundation (FCECON), using Samsung® gear VR virtual reality glasses and Samsung® smart watch.
  Interventions: Device: Case group
- Active Control Group (Active Comparator): The active control group will watch a 7-minute mindfulness meditation video presented via cell phone with image and sound in the office of the Oncology Control Center Foundation (FCECON), using a Samsung® smart watch.
  Interventions: Behavioral: Active control group
- Passive Control Group (Active Comparator): The passive control group will perform meditation breathing exercises based on instructions and through an audio played from the health professional for 4 minutes in the office of the Oncology Control Center Foundation (FCECON), using a Samsung® smart watch.
  Interventions: Behavioral: Passive control group

INTERVENTIONS:
Device: Case group — Meditation will be taught through a video played on a Samsung® gear VR virtual reality glasses with monitoring of the patient's vital signs by the Samsung® smart watch to promote better quality of life and control cancer pain in patients treated at the Pain Therapy and Palliative Care Service.
  Arms: Case Group
Behavioral: Active control group — Meditation will be taught through a video played on a Samsung® cell phone with monitoring of the patient's vital signs by the Samsung® smart watch to promote better quality of life and control cancer pain in patients treated at the Pain Therapy and Palliative Care Service.
  Arms: Active Control Group
Behavioral: Passive control group — Meditation will be taught through a audio played on a Samsung® cell phone with monitoring of the patient's vital signs by the Samsung® smart watch to promote better quality of life and control cancer pain in patients treated at the Pain Therapy and Palliative Care Service.
  Arms: Passive Control Group

SUMMARY:
Cancer is a disabling, challenging and growing global disease. Although early diagnosis and adequate treatment of oncological disease have been developing rapidly, a large part of the population remains without access to specialized services and routinely evolve to symptoms and sequelae with uncontrolled pain, worse quality of life and suffering. Complementary therapies to control pain and improve the well-being of cancer patients are fundamental tools of integrative oncology medicine. This study proposes to use immersive virtual reality to encourage cancer patients to carry out the regular practice of meditation, as an effective tool in pain management and in the search for a better quality of life, based on a structured intervention that encourages autonomy as important part of your treatment. Two studies will be carried out at the Pain Therapy and Palliative Care Service of the Amazonas State Oncology Control Center Foundation (FCECON). Study 1 will be a cross-sectional study to describe the variables associated with the diagnosis and treatment of patients' pain and Study 2 will be a Randomized Controlled Trial that will analyze the impact of an intervention performed with meditation through immersive virtual reality for pain relief. pain in these patients. It is expected that the regular practice of meditation through immersive virtual reality will promote pain relief and improve the quality of life of cancer pain patients.

DETAILED DESCRIPTION:
This is a prospective, experimental, longitudinal study of the randomized controlled trial (RCT) type, carried out in three stages. Randomization will be carried out entirely using a specific application called Randomizer ® for Clinical Trial Lite. The defined sample was 39 participants per group. This would mean a total of 117 participants, divided into 3 groups of 39 participants each. Furthermore, considering the possibility of loss to follow-up, 12% was added to the final figure of 39 participants, due to the possibility of loss to follow-up, giving a final sample of 129 participants, divided into 3 groups: Experimental group; Passive control group and Active control group, with 43 participants in each group. At moment 1 (M1) all the patients will answer the sociodemographic and clinical questionnaire, and the other Quality of Life, Psychological Morbidity, pain scale and symptom scale instruments, after which they will perform the meditation used in the group to which they were randomly assigned, in the experimental case group (Group A) a 7-minute immersive virtual reality video of mindfulness meditation with image and sound in a comfortable chair in the office of the Oncology Control Center Foundation (FCECON), using Samsung® gear virtual reality (VR) glasses and Samsung® smartwatch; in the active control group (Group B) a 7-minute video of mindfulness meditation on a cell phone with image and sound in a comfortable chair in the office of the Oncology Control Center Foundation (FCECON), using Samsung® smart watch; and in the passive control group (Group C) breathing exercises based on instructions from the health professional for 4 minutes in a comfortable chair in the office of the Oncology Control Center Foundation (FCECON), using Samsung® smart watch. After watching the video, all patients will answer the 4 Quality of Life, Psychological Morbidity, pain scale and symptom scale instruments and will receive instructions on how to perform the meditation, using a free app that offers mindfulness meditation videos for offline use with images and sound for 3 minutes three times for 4 weeks in a home environment. They will receive Short Message Service (SMS) alerts on their cell phones to remind them to do the video-guided home meditation on Mondays, Wednesdays and Fridays between 9am and 10am. A printed form will be given to each patient with the dates of the meditation to mark their satisfaction with the meditation by classifying it as totally dissatisfied - I hated it, dissatisfied - I didn't like it, indifferent, satisfied - I liked it or totally satisfied - I loved it. All the previous steps will be repeated in Moment 2 (M2), 4 weeks after Moment 1 (about 1 month), and in Moment 3 (M3): 8 weeks after Moment 1 (about 2 months). All patients, regardless of group, will be taught by different means to practice guided meditation regularly and will use the Samsung Smart watch Galaxy Watch6 LTE 44mm Super Active Matrix Organic Light Emitting Diode (AMOLED) Screen 1.47, Graphite, exclusively during the interview and meditation, handled by the researcher, at the Pain Therapy and Palliative Care Service of the Oncology Control Center Foundation (FCECON), at the three moments of the research. This watch has the following devices and capabilities: "BioActive Sensor - Optical Heartbeat, Electrocardiogram and Bioelectrical Impedance Analysis, in addition to the customizable heart rate zone, the Oximeter, Fall Detection and Emergency Call, and sleep quality monitoring". And it will be used to track quantitative variables: heart rate and blood oxygen saturation. It will also allow the patient to be monitored using the Brazilian version of the Distress Thermometer and Problem List from the National Comprehensive Cancer Network (NCCN), which is a free resource that identifies and addresses unpleasant experiences that can make it more difficult to deal with cancer, its symptoms or treatment. Finally, it will also be possible to use the smart watch to answer the visual pain scale for audio feedback. All participants will use their own Android cell phone with the functions installed for the use of the smartwatch and it will capture body movement data by acceleration signals, location with anonymized global positioning system (GPS) data, encrypted speech. The mobile questionnaire app, the visual pain scale and the Brazilian version of the Distress Thermometer and Problem List from the National Comprehensive Cancer Network (NCCN) - will be installed.

ELIGIBILITY:
Inclusion Criteria:

* Be followed up at the Pain Therapy and Palliative Care Service (STDCP) to control symptoms resulting from any type of cancer at any stage;
* Have a diagnosis of chronic pain, recorded in the medical records.
* Be between 18 and 75 years old on the date of the first collection;
* Be able to understand Portuguese (read and write);
* Have normal vision and hearing;
* Have a cell phone with an Android system;
* Be able to make head movements and have sufficient motor control to make body movements;
* Agree to take part in the study and sign the Informed Consent Form (ICF).

Exclusion Criteria:

* Indigenous patients (due to cultural and linguistic peculiarities and special legislation);
* Patients with records of serious psychiatric illnesses (DSM-5 - Diagnostic and Statistical Manual of Mental Disorders - schizophrenia, schizotypal disorders, delusional disorders, borderline and dementias);
* Impairment of the ability to understand or communicate based on the researcher's assessment;
* Report of discomfort with the use of Immersive Virtual Reality;
* Progression of the disease with limitation in maintaining the proposed regular outpatient visits;
* Patients with brain tumors, brain metastases or a previous history of seizures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (Reduced version) | six months
  It has a body schema, in which the patient can mark the location of the pain, as well as 8 questions relating to pain intensity, on a scale of 0 to 10, the higher the score on the inventory, the worse the pain intensity.
McGill Quality of Life Questionnaire | six months
  Made up of 16 items, divided into domains: physical well-being, psychological well-being, existential well-being, support and physical symptoms. It has a single-item scale that measures overall quality of life, which is not included in the score, but is used to compare scores. It also has an open question for the patient to name the things that have had the greatest effect on their quality of life. The scale has eleven points from 0 to 10, and the higher the final score, the better the quality of life.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | six months
  A 14-item instrument with two sub-scales, anxiety and depression, with seven items each to assess depression and anxiety. The score for each item can vary from zero to three, with a maximum score of 21 points for each sub-scale (anxiety and depression). Patients with no anxiety/depression are considered to score from 0 to 8, and ≥ 9 have anxiety/depression.
The Edmonton Symptom Assessment Scale (ESAS) | six months
  The ESAS is a simple, self-reported questionnaire designed to indicate objective and subjective symptoms. On this scale, the patient or their caregiver/family member assigns a score from 0 to 10 for each symptom, with 0 being the absence and 10 the greatest intensity of the symptom.
The National Comprehensive Cancer Network® (NCCN) Distress Thermometer | six months
  The National Comprehensive Cancer Network® (NCCN) Distress Thermometer will be applied as a questionnaire during the 3 moments. It is a translated and validated NCCN tool used to measure the "temperature" of the mental health of people with cancer. The Brazilian version of the NCCN Distress Thermometer and Problem List.

CONTACTS AND LOCATIONS:
Overall Officials: Emily S Montarroyos, Principal Investigator — Fundação Centro de Controle de Oncologia do Estado do Amazonas (FCECON)
Locations (1):
- Fundação Centro de Controle de Oncologia do Estado do Amazonas - FCECON, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swami M, Case AA. Effective Palliative Care: What Is Involved? Oncology (Williston Park). 2018 Apr 15;32(4):180-4. PMID 29684230
- [Background] Sheinfeld Gorin S, Krebs P, Badr H, Janke EA, Jim HS, Spring B, Mohr DC, Berendsen MA, Jacobsen PB. Meta-analysis of psychosocial interventions to reduce pain in patients with cancer. J Clin Oncol. 2012 Feb 10;30(5):539-47. doi: 10.1200/JCO.2011.37.0437. Epub 2012 Jan 17. PMID 22253460
- [Background] Lyman GH, Greenlee H, Bohlke K, Bao T, DeMichele AM, Deng GE, Fouladbakhsh JM, Gil B, Hershman DL, Mansfield S, Mussallem DM, Mustian KM, Price E, Rafte S, Cohen L. Integrative Therapies During and After Breast Cancer Treatment: ASCO Endorsement of the SIO Clinical Practice Guideline. J Clin Oncol. 2018 Sep 1;36(25):2647-2655. doi: 10.1200/JCO.2018.79.2721. Epub 2018 Jun 11. PMID 29889605
- [Background] Mao JJ, Ismaila N, Bao T, Barton D, Ben-Arye E, Garland EL, Greenlee H, Leblanc T, Lee RT, Lopez AM, Loprinzi C, Lyman GH, MacLeod J, Master VA, Ramchandran K, Wagner LI, Walker EM, Bruner DW, Witt CM, Bruera E. Integrative Medicine for Pain Management in Oncology: Society for Integrative Oncology-ASCO Guideline. J Clin Oncol. 2022 Dec 1;40(34):3998-4024. doi: 10.1200/JCO.22.01357. Epub 2022 Sep 19. PMID 36122322
- [Background] Aisenberg-Shafran D, Shturm L. The effects of mindfulness meditation versus CBT for anxiety on emotional distress and attitudes toward seeking mental health treatment: a semi-randomized trial. Sci Rep. 2022 Nov 16;12(1):19711. doi: 10.1038/s41598-022-24256-9. PMID 36385638
- [Background] Deng G. Integrative Medicine Therapies for Pain Management in Cancer Patients. Cancer J. 2019 Sep/Oct;25(5):343-348. doi: 10.1097/PPO.0000000000000399. PMID 31567462
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Mo J, Vickerstaff V, Minton O, Tavabie S, Taubert M, Stone P, White N. How effective is virtual reality technology in palliative care? A systematic review and meta-analysis. Palliat Med. 2022 Jul;36(7):1047-1058. doi: 10.1177/02692163221099584. Epub 2022 May 30. PMID 35635018
- [Background] Mao JJ, Pillai GG, Andrade CJ, Ligibel JA, Basu P, Cohen L, Khan IA, Mustian KM, Puthiyedath R, Dhiman KS, Lao L, Ghelman R, Caceres Guido P, Lopez G, Gallego-Perez DF, Salicrup LA. Integrative oncology: Addressing the global challenges of cancer prevention and treatment. CA Cancer J Clin. 2022 Mar;72(2):144-164. doi: 10.3322/caac.21706. Epub 2021 Nov 9. PMID 34751943
- [Background] Latte-Naor S, Mao JJ. Putting Integrative Oncology Into Practice: Concepts and Approaches. J Oncol Pract. 2019 Jan;15(1):7-14. doi: 10.1200/JOP.18.00554. PMID 30629900
- [Background] Bao T, Greenlee H, Lopez AM, Kadro ZO, Lopez G, Carlson LE. How to Make Evidence-Based Integrative Medicine a Part of Everyday Oncology Practice. Am Soc Clin Oncol Educ Book. 2023 May;43:e389830. doi: 10.1200/EDBK_389830. PMID 37200595
- [Background] Austin PD, Siddall PJ, Lovell MR. Feasibility and acceptability of virtual reality for cancer pain in people receiving palliative care: a randomised cross-over study. Support Care Cancer. 2022 May;30(5):3995-4005. doi: 10.1007/s00520-022-06824-x. Epub 2022 Jan 21. PMID 35064330
- [Background] Guenther M, Gorlich D, Bernhardt F, Pogatzki-Zahn E, Dasch B, Krueger J, Lenz P. Virtual reality reduces pain in palliative care-A feasibility trial. BMC Palliat Care. 2022 Oct 5;21(1):169. doi: 10.1186/s12904-022-01058-4. PMID 36195865
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113
- [Background] Ferreira KA, Teixeira MJ, Mendonza TR, Cleeland CS. Validation of brief pain inventory to Brazilian patients with pain. Support Care Cancer. 2011 Apr;19(4):505-11. doi: 10.1007/s00520-010-0844-7. Epub 2010 Mar 10. PMID 20221641
- [Background] Seiler A, Schettle M, Amann M, Gaertner S, Wicki S, Christ SM, Theile G, Feuz M, Hertler C, Blum D. Virtual Reality Therapy in Palliative Care: A Case Series. J Palliat Care. 2026 Jan;41(1):19-27. doi: 10.1177/08258597221086767. Epub 2022 Mar 16. PMID 35293818
- [Derived] Montarroyos ES, Lima S, Barreto R, Moyses R, Cardenas LZ. Integrating Immersive Virtual Reality Meditation into Palliative Oncology: A Randomized Trial Protocol for Evaluating Pain Relief and Quality of Life. Healthcare (Basel). 2026 Jan 21;14(2):266. doi: 10.3390/healthcare14020266. PMID 41595402
- See also: Ministry of Health. National Cancer Institute. Estimates of Cancer Incidence in Brazil. Estimates 2023. Rio de Janeiro: INCA, 2022. — https://www.inca.gov.br/sites/ufu.sti.inca.local/files/media/document/dieta_nutricao_atividade_fisica_e_cancer_resumo_do_terceiro_relatorio_de_especialistas_com_uma_perspectiva_brasileira.pdf
- See also: National Comprehensive Cancer Network. A tool translated from the NCCN measures the "temperature" of the mental health of people with cancer. — https://www.prnewswire.com/news-releases